CLINICAL TRIAL: NCT00040729
Title: Retrospective Analysis Of Promoter Polymorphism Of UGT1A1 Gene In Cancer Patients Enrolled On Clinical Trials With Flavopiridol At National Cancer Institute To Assess The Pharmacokinetics And Pharmacodynamics Of Flavopiridol
Brief Title: Genetic Study of Patients Previously Treated With Flavopiridol on Clinical Trial NCI-97-C-0171C
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000069394; NCI-02-C-0161
Record Dates: First submitted 2002-07-08; First posted 2003-06-26 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2003-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

INTERVENTIONS:
Genetic: mutation analysis

SUMMARY:
RATIONALE: Genetic testing for a specific enzyme may help doctors determine whether side effects from or response to chemotherapy are related to a person's genetic makeup.

PURPOSE: Genetic trial to determine whether different forms of the UGT1A1 gene are related to the body's ability to break down drugs and to the gastrointestinal side effects seen in patients previously treated with flavopiridol.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the relationship between UGT1A1 genotypes and drug pharmacokinetics and occurrence of gastrointestinal toxicity in cancer patients previously treated with flavopiridol on protocol NCI-97-C-0171C.

OUTLINE: Genomic DNA from pre-existing samples of serum or plasma from each patient is analyzed for UGT1A1 gene by polymerase chain reaction and DNA sequencing. Results are then analyzed for a possible association between UGT1A1 genotypic variation and susceptibility to flavopiridol.

Patients do not receive the results of the genetic testing, and the results do not influence the type or duration of treatment.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cancer patients previously treated with flavopiridol on protocol NCI-97-C-0171C

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-03

CONTACTS AND LOCATIONS:
Overall Officials: William D. Figg, PharmD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States